CLINICAL TRIAL: NCT01311440
Title: Modified Atkins Diet Treatment for Adults With Drug-resistant Epilepsy - a Controlled, Randomized Trial
Brief Title: Modified Atkins Diet Treatment for Adults With Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnhild Kverneland, Registered Nutritionist, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/2326 (REK)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy; Focal Epilepsy; Generalized Epilepsy
Keywords: RCT; modified Atkins diet; epilepsy; adults; ketogenic diet
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Epilepsy, Generalized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Atkins diet treatment (Experimental): 12 weeks of Modified Atkins diet treatment, recording seizures
  Interventions: Other: Modified Atkins diet treatment
- No intervention (No Intervention): 12 weeks seizure record

INTERVENTIONS:
Other: Modified Atkins diet treatment — Eat a diet containing 16 grams of carbohydrates per day, maximize on fat. Assure sufficient intake of micronutrients.
  Arms: Modified Atkins diet treatment

SUMMARY:
In Oslo University Hospital, department of complex epilepsy, offer ketogenic diet to treat children with medically intractable epilepsy. From 2009 we added modified Atkins diet as a treatment option for children up to 18 years.

We now initiate an open, prospective, randomized and controlled study with the aim to test the efficacy of treatment with modified Atkins diet in adults with focal and generalized epilepsy diagnoses, in order to evaluate whether this treatment should be offered to patients on a permanent basis.

DETAILED DESCRIPTION:
Poorly controlled epilepsy in adults affects health and quality of life in many ways. Within this heterogenous population there are individuals who are motivated for a very strict diet in order to reduce seizures.

Among adults with epilepsy 75 - 80 % are diagnosed with focal epilepsy, while 20 - 25 % have generalized onset of seizures.

We plan to include 92 patients with focal epilepsy diagnosis. Those are randomized into diet and control groups.

During the inclusion period we also treat patients with generalized epilepsy that qualify for participation, but these are not to be randomized, rather they will follow the diet group course. We assume 18 - 23 patients with generalized epilepsy will be included in the project.

ELIGIBILITY:
Inclusion Criteria:

* Focal or generalized epilepsy diagnosis
* More than 3 recordable seizures per month
* BMI > 18,5
* Not responded to at least three 3 AEDs
* 16 years or older
* Motivated to complete the diet after thorough information
* Capable of recording seizures
* Capable of preparing the diet

Exclusion Criteria:

* Hypercholesterolemia, cardiovascular disease or kidney disease
* Been on modified Atkins diet for more than one week during the last year
* Status epilepticus last six months
* epilepsy surgery or VNS implant last year
* 4 weeks continuous seizure freedom last 2 months
* PNES seizures
* other disease where dietary treatment is contraindicated
* usage of drugs or supplements that may interfere with diet or AED
* being pregnant or planning pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | 12 weeks
  All participants record detailed seizure records for 12 weeks prior to the control/diet period. The diet group participants are subsequently treated with modified Atkins diet for 12 weeks, while the control group continue their normal diet and record seizures for another 12 weeks. Seizure records for each participant before and during intervention are compared.

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
Change in standard 3-hrs EEG | 12 weeks
Change in life quality measured by validated questionnaire | 12 weeks
Change in various blood and serum measures | 12 weeks
Change in executive functions measured with validated questionnaire | 12 weeks
Change in seizure strength and severity measured by validated questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Otto Nakken, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, The national Centre for epilepsy, Sandvika, Bærum Postterminal, Norway

IPD SHARING:
Plan to Share IPD: Undecided